CLINICAL TRIAL: NCT05656976
Title: Efficacy of Offering a Self-sampling Device by the General Practitioner to Reach Women Underscreened in the Routine Cervical Cancer Screening Program Compared to Sending Reminder Letters by the Screening Organization
Brief Title: Efficacy of Offering a Self-sampling Device by the GP to Reach Underscreened Women
Acronym: ESSAG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Ghent (Other)
Collaborators: Kom Op Tegen Kanker (Other); Sciensano (Other Government); Centrum voor Kankeropsporing (Unknown); Belgian Cancer Registry (Other); KU Leuven (Other); Vrije Universiteit Brussel (Other); Universiteit Antwerpen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: ONZ-2022-0250
Record Dates: First submitted 2022-11-23; First posted 2022-12-20 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Cervical Cancer
Keywords: Prevention; Screening
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial (RCT)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- A Self sampling device (SSD) provided by the general practitioner (GP) (Experimental): A self sampling device will be provided by the GP.
  Interventions: Other: Provision of self sampling device by the GP
- B Self sampling device provided by letter (Experimental): A self sampling device will be provided by letter.
  Interventions: Other: Provision of self sampling device by letter
- C (control arm) Recommendation letter (No Intervention): Following the usual care procedure, a random sample of 1125 Flemish women who meet the same inclusion criteria as in arm A and B and are not included in one of the latter arms is drawn by "Centrum voor Kankeropsporing" (CvKO) from Heracles, the database of the Flemish screening program.

INTERVENTIONS:
Other: Provision of self sampling device by the GP — In a group of 45 GP practices, over a course of 9 months, all long-term unscreened women with a GMD will be addressed by their GP when they consult for any reason. The GP will discuss the pros and cons of screening for cervical cancer, the various options for screening for cervical cancer including the possibility of using a SSD. For this, the GP can use on accessible brochure and video materials. After the woman agrees, she is given a self-taking kit that she can use when and where it suits her and send it to the lab with the prepaid envelope. The woman is informed of the result of the Human Papilloma Virus test result by her GP according to the usual way in the practice (e.g. via letter, by phone or during the next consultation).
  Arms: A Self sampling device (SSD) provided by the general practitioner (GP)
Other: Provision of self sampling device by letter — In the second arm, a second group of 45 GP practices in Flanders will be recruited. With the intervention of the Centre for Cancer Prevention (Flanders), 25 at randomly selected long-term unscreened women with a Global Medical Form (in dutch: 'Globaal Medisch Dossier, GMD) in one of these practices will receive an envelope containing a letter of invitation from their GP for cervical cancer screening, a brochure with the advantages and disadvantages of cervical cancer screening and more specifically the use of a self-taking kit, and a self-taking kit. If the woman wishes, she can use the kit when and where it suits her and send it to the lab with the pre-paid envelope. As in arm A, the woman will be informed of the Human Papilloma Virus test result by her GP according to the usual way in the practice (e.g., by letter, by phone or during the next consultation). All women will receive a study-related reminder letter after 4 months.
  Arms: B Self sampling device provided by letter

SUMMARY:
The ESSAG trial invests the impact of offering a free self-sampling device (SSD) on the cervical cancer screening rate of underscreened women. This study is aimed at women between the age of 31 and 65 who did not have a smear taken during the last 6 years. In order to assess the effect of a) providing the SSD, and b) the intervention of the general practitioner (GP) (either face-to-face, either by sending the SSD by letter), a randomized control trial is set up with three arms. The ESSAG trial evolves from a collaboration between Universiteit Gent and Vrije Universiteit Brussel, Katholieke Universiteit Leuven, Universiteit Antwerpen, Sciensano, het Centrum voor Kankeropsporing en het Belgisch Kankerregister, and is funded by "Kom Op Tegen Kanker".

ELIGIBILITY:
Inclusion Criteria:

* women between 31-64 years old
* living in Flanders
* eligible for the Flemish actions with regard to population screening
* without a smear registered in the Belgian Cancer Registry in the last 6 years
* registered as GMD patient in one of the participating GP practices

Exclusion Criteria:

* hysterectomy
* pregnancy
* (past) diagnosis of cervical cancer

Ages: 31 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 3375 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Response rate | Up to 6 months
  Age-standardised response rates in each arm and the differences between arms will be calculated, in a per protocol (PP) and intention-to-treat (ITT) analysis.
  As the goal is to reveal to what extent the respective approach (providing a self sampling device (SSD) with different levels of general practitioner (GP) involvement) succeeds in reaching vulnerable women, analyses will take into account a comprehensive list of covariates by logistic regression accounting for cluster effects. These covariates include trial arm, GP-office characteristics, as well as demographic information of the patient on origin and socio-economical background provided by the "Kruispuntbank voor Sociale Zekerheid (KSZ)".

SECONDARY OUTCOMES:
Participation rate | Up to 9 months
  The participation rate will be calculated from arm A to answer questions at public health level, i.e. the population effect of the intervention by GP's on increasing cervical cancer screening coverage in underscreened women.
  For participation rate, the denominator are all women who belong to the target group for that specific GP-office (women between 31-64y, not screened within 6y, etc).
Cost-effectiveness analysis | Up to 15 months
  A cost-effectiveness analysis will also be performed, addressing the additional number of women screened per 1,000€ in interventions A and B versus control intervention C.
Feasibility analysis (semi-structured interviews with GP's) | Up to 4 months after the intervention in their practice
  In order to explore the potential roll-out of the study within the Flemish screening programme, the investigators will also perform a feasibility study. Through interviews with 20-30 GPs who participated in arm A, a feasibility analysis will reveal the strengths and pitfalls of the intervention.
Response rate (follow-up cytology test) | Up to 3 months
  Although this study is not powered for inter-arm differences in follow-up after an abnormal screening test result, compliance analysis will be performed with the following indicators: screen-test positivity rates, proportion with invalid screen-test results, proportion of screen-test positives that have the foreseen follow-up tests.

CONTACTS AND LOCATIONS:
Overall Officials: Kaatje Van Roy, Principal Investigator — University Ghent
Locations (1):
- Ghent University, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gezels E, Van Roy K, Arbyn M, Coursier P, Devroey D, Martens P, Simoens C, Vaes B, Van Herck K, Vankrunkelsven P, Verhoeven V, Willems S. The ESSAG-trial protocol: A randomized controlled trial evaluating the efficacy of offering a self-sampling kit by the GP to reach women underscreened in the routine cervical cancer screening program. Contemp Clin Trials. 2024 Sep;144:107617. doi: 10.1016/j.cct.2024.107617. Epub 2024 Jul 6. PMID 38977179